CLINICAL TRIAL: NCT03127176
Title: Dysbiosis in Bipolar Disorder: MicrObiota Bipolar Study
Brief Title: Dysbiosis in Bipolar Disorder
Acronym: MOB
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Iria Grande, Principal Investigator, Hospital Clinic of Barcelona
Other Study IDs: PI 16/00187
Record Dates: First submitted 2017-03-29; First posted 2017-04-25 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample

GROUPS / COHORTS (3):
- BD with cognitive impairment: This group will include euthymic patients with bipolar disorder type I or II (YMRS<6 and HMDRS<8) and cognitive impairment.
  Intervention: Genome sequencing of fecal samples
  Interventions: Other: Genome sequencing of fecal samples
- BD without cognitive impairment: This group will include euthymic patients with bipolar disorder type I or II (YMRS<6 and HMDRS<8) without cognitive impairment.
  Intervention: Genome sequencing of fecal samples
  Interventions: Other: Genome sequencing of fecal samples
- Control group: This group will include healthy volunteers. Intervention: Genome sequencing of fecal samples
  Interventions: Other: Genome sequencing of fecal samples

INTERVENTIONS:
Other: Genome sequencing of fecal samples — Fecal samples will be collected and then frozen in the morning pre-prandial after having fasted overnight. DNA will be separated and stored at -80°C in our center (Biobanc) until assayed. Sequencing will be performed with the most appropriate platform.

SUMMARY:
The gut microbiota is a complex community comprising around 10^14 bacteria that live in the gut lumen. The imbalance of the normal structure and function of the microbiota, defined as dysbiosis, has been related to a wide diversity of pathologies, including mental health disorders. However, clinical evidence of the relationship between microbiota and mood disorders is lacking. The aim of this project is to examine the possible relationship of gut dysbiosis and the diagnosis of bipolar disorder (BD), of gut dysbiosis and mood relapses and of gut dysbiosis and cognitive impairment in bipolar patients.

DETAILED DESCRIPTION:
A prospective longitudinal study will be carried out with three groups of patients: a group of euthymic bipolar I or II patients without cognitive impairment (n=50), a second group of euthymic bipolar I or II patients with cognitive impairment (n=50) and a control group of healthy volunteers (n=50). Cognitive impairment will be defined as performance in any test of a domain below 2 standard deviations or more from the mean of normative data of each test assessed in the control group. Subjects will be recruited in the Hospital Clinic of Barcelona. At baseline clinical variables and diet patterns (ROME III) will be collected and neuropsychological performance (WCST, FAS, Stroop Colour-Word Interference test, TMT, WAIS-III, CVLT-II) and functionality (FAST) will be assessed. All subjects will be reassessed at 12 months follow-up. The mood state and possible affective relapses will be evaluated and treatments will be registered. All patients will receive standard psychiatric care according to international guidelines on bipolar disorders. Fecal samples will be collected and then frozen in the morning pre-prandial after having fasted overnight. DNA will be separated and stored at -80°C until assayed. Sequencing will be performed on an Illumina MiSeqTM platform. Statistical analysis will be performed with the latest existing version of the SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Diagnosis of bipolar disorder type I or II according to DSM-IV criteria (SCID);
  * Age between 18-55 years;
  * Euthymia (YMRS<6 and HMDRS<8) for at least 3 months;
  * Signed informed consent.
* Healthy controls:

  * No psychiatric diagnosis (SCID);
  * Age between 18-55 years; euthymia (YMRS<6 and HMDRS<8);
  * Signed informed consent.

Exclusion Criteria:

* Use of any type of antibiotics, antifungals or pro/prebiotics within at least one month prior to recruitment;
* IQ<85;
* Neurological illness;
* Stomach/gut problems;
* Current diagnosis of substance abuse or dependence according to DSM-IV criteria (SCID);
* Electroconvulsive therapy in the last year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with BD will be recruited in the Bipolar Unit outpatient clinic in the Hospital Clinic of Barcelona. Healthy volunteers will be selected from the community.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Composition of the gut microbiota. | 12 months
  To determine if patients diagnosed with BD present gut dysbiosis compared to controls through genome sequencing of fecal samples.

SECONDARY OUTCOMES:
Composition of the gut microbiota according to mood state. | 12 months
  Gut dysbiosis will be determined according to mood state, assessed using clinical evaluation.
Composition of the gut microbiota according to cognitive state. | 12 months
  Gut dysbiosis will be determined according to cognitive state, assessed using a pre-defined neuropsychological battery.

CONTACTS AND LOCATIONS:
Overall Officials: Iria Grande, MD, PhD, Principal Investigator — Bipolar Disorders Unit, Hospital Clinic, Institute of Neurosciences, University of Barcelona, IDIBAPS, CIBERSAM
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided